CLINICAL TRIAL: NCT05687071
Title: A Multicenter, Open-label, Uncontrolled, Long-term Trial to Assess the Safety and Efficacy of ETC-1002 in Patients With Hyper-LDL Cholesterolemia
Brief Title: A Long-term Trial of ETC-1002 in Patients With Hyper-LDL Cholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 346-102-00003
Record Dates: First submitted 2023-01-04; First posted 2023-01-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hyper-low-density Lipoprotein (LDL) Cholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ETC-1002 180mg (Experimental)
  Interventions: Drug: 180mg of ETC-1002(bempedoic acid)

INTERVENTIONS:
Drug: 180mg of ETC-1002(bempedoic acid) — 180mg, tablet, once daily, for 52 weeks

SUMMARY:
A Multicenter, Open-label Study to assess the safety and efficacy of ETC-1002 at 180 mg administered for 52 weeks in patients with hyper-LDL cholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Patients with inadequate response to statins or who have difficulty in treatment with statins as defined below [Inadequate response to statins] Patients with hyper-LDL cholesterolemia who are currently taking or have previously taken statins[and other lipid-modifying therapies(LMTs) if needed] and cannot achieve the lipid management goals of LDL-C [Difficulty in treatment with statins] Patients with hyper-LDL cholesterolemia for whom safety problems have occurred while taking at least one type of statin, and who experienced resolution of the problems after discontinuation or dose reduction, or of those patients who have a history of statin administration and who are judged to have concerns of safety problems associated with the administration or dose increase of statins and who cannot achieve the lipid management goals of LDL-C. Patients must be on the lowest or under the dosage of the approved dose of statin and/or on stable LMT(s).
* Patients with fasting TG levels of <400 mg/dL at screening
* Other protocol specific inclusion criteria may apply

Exclusion Criteria:

* Females who are pregnant or breast-feeding or who have a positive pregnancy test (urine) result at screening or baseline visits
* Patients with homozygous familial hypercholesterolemia (HoFH)
* Patients who currently have or who have had within the past 3 months prior to screening any cardiovascular diseases, or those who have developed any cardiovascular diseases during the screening
* Uncontrolled hypertension, defined as sitting systolic blood pressure after resting 5 minutes of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg at screening
* Patients with uncontrolled and serious hematologic or coagulation disorders or with hemoglobin of <10.0 g/dL at screening
* Patients with uncontrolled diabetes with HbA1c of ≥9% at screening
* Patients with uncontrolled hypothyroidism with thyroid-stimulating hormone (TSH) of >1.5 × ULN at screening
* Patients with liver disease or dysfunction, including:

  * Positive serology for hepatitis B surface antigen (HBsAg) or a positive hepatitis C virus (HCV) antibody test at screening
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) of ≥3 × ULN or total bilirubin of ≥2 × ULN at screening
* Patients with creatine kinase (CK) of >3 × ULN at screening
* Patients with a history or current renal dysfunction, nephritic syndrome, or nephritis, and with estimated glomerular filtration rate (eGFR) of ≤30 mL/min/1.73 m2 at screening
* Other protocol specific exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-11-02 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Treatment-Emergent Adverse Events (TEAEs) | From baseline to week 52
Percent change in low-density lipoprotein cholesterol (LDL-C) from baseline to Week 52 | Baseline, week52

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Rinku General Medical Center, Izumisano, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.